CLINICAL TRIAL: NCT01655069
Title: An Open-Label, Long-Term Extension, Multi-center, Sequential Dose Titration Study to Assess Safety and Efficacy of Solifenacin Succinate Suspension in Pediatric Subjects With Overactive Bladder (OAB)
Brief Title: A Study to Investigate How Safe and Effective Solifenacin Solution is in Treating Children/Adolescents With Symptoms of Overactive Bladder (OAB) Who Completed Study 905-CL-076
Acronym: LEOPARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 905-CL-077; 2011-002047-10 (EudraCT Number)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive bladder (OAB); Solifenacin succinate suspension; Phase 3; Pediatric
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Children Treated with Placebo in 905-CL-076 (Experimental): Male and female children aged 5 to less than 12 years old who received placebo in Study 905-CL-076 and received open-label solifenacin once daily in this study. The mean time on study drug in this study was 247.9 days in children.
  Interventions: Drug: Solifenacin succinate suspension
- Children Treated with Solifenacin in 905-CL-076 (Experimental): Male and female children aged 5 to less than 12 years old who received solifenacin in Study 905-CL-076 and received open-label solifenacin once daily in this study. The mean time on study drug in this study was 247.9 days in children.
  Interventions: Drug: Solifenacin succinate suspension
- Adolescents Treated with Placebo in 905-CL-076 (Experimental): Male and female adolescents aged 12 to less than 18 years old who received placebo in Study 905-CL-076 and received open-label solifenacin once daily in this study. The mean time on study drug in this study was 240.1 days in adolescents.
  Interventions: Drug: Solifenacin succinate suspension
- Adolescents Treated with Solifenacin in 905-CL-076 (Experimental): Male and female adolescents aged 12 to less than 18 years old who received solifenacin in Study 905- CL-076 and received open-label solifenacin once daily in this study. The mean time on study drug in this study was 240.1 days in adolescents.
  Interventions: Drug: Solifenacin succinate suspension

INTERVENTIONS:
Drug: Solifenacin succinate suspension — Oral suspension
  Other Names: YM905; solifenacin succinate

SUMMARY:
This was a 40-week study to investigate how safe and effective solifenacin solution was in treating children or adolescents with symptoms of overactive bladder (OAB), who completed study 905-CL-076 (NCT01565707).

DETAILED DESCRIPTION:
There was a titration period of up to 12 weeks during which the participants would be up or down-titrated based on a combination of efficacy and safety parameters followed by a fixed dose period during which no dose adjustments were allowed. Participants completed a 7-day patient diary prior to every visit (start of 905-CL-076 to end of 905-CL-077, 14 visits). The first visit of this study (905-CL-077) was combined with the last visit of the 4-month study 905-CL-076. At each visit, the participant was required to undertake a number of assessments or examinations to determine whether it is safe for him/her to take part or to continue to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has met the inclusion criteria of study 905-CL-076 and completed study 905-CL-076

Exclusion Criteria:

* Subject has failed the exclusion criteria of study 905-CL-076

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2014-10-08 (Actual); Study Completion 2014-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (39):
- Site: 1006, Shreveport, Louisiana, United States
- Belgium (7):
  - Site: 3202, Antwerp
  - Site: 3209, Antwerp
  - Site: 3208, Charleroi
  - Site: 3201, Ghent
  - Site: 3203, Ghent
  - Site: 3204, Kortrijk
  - Site: 3205, Leuven
- Brazil (2):
  - Site: 5507, Campinas
  - Site: 5506, Curitiba
- Site: 1001, Québec, Canada
- Denmark (4):
  - Site: 4503, Aalborg
  - Site: 4501, Aarhus N
  - Site: 4502, Kolding
  - Site: 4504, Køge
- Mexico (2):
  - Site: 5202, Mexico City
  - Site: 5205, Mexico City
- Site: 4701, Bergen, Norway
- Site: 6301, Quezon City, Philippines
- Poland (4):
  - Site: 4805, Gdansk
  - Site: 4803, Gdansk
  - Site: 4804, Lubin
  - Site: 4801, Warsaw
- Serbia and Montenegro (2):
  - Site: 3810, Belgrade
  - Site: 3812, Novi Sad
- Site: 2703, Cape Town, South Africa
- South Korea (4):
  - Site: 8203, Daegu
  - Site: 8206, Incheon
  - Site: 8207, Seoul
  - Site: 8202, Seoul
- Sweden (4):
  - Site: 4606, Gothenburg
  - Site: 4603, Skövde
  - Site: 4602, Stockholm
  - Site: 4605, Umeå
- Turkey (Türkiye) (2):
  - Site: 9001, Ankara
  - Site: 9002, Izmir
- Site: 3854, Kharkiv, Ukraine
- United Kingdom (2):
  - Site: 4403, Leeds
  - Site: 4401, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-002047-10/results
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this study were children (5 to less than 12 years old) and adolescents (12 to less than 18 years old) with overactive bladder (OAB), who completed the 2-week placebo run-in period and 12-week treatment period of Study 905-CL-076 (NCT01565707).
Pre-assignment Details: Children and adolescents with OAB, who completed study 905-CL-076, consented to enter this study and fulfilled all the eligibility criteria were enrolled at Week 12/13 (2-3 days after last dose was received during the 905-CL-076 study). The age of participant at informed consent signing in 905-CL-076 determined the age group in this study.
Period: Overall Study
Arm/Group | Children Treated With Placebo in 905-CL-076 | Children Treated With Solifenacin in 905-CL-076 | Adolescents Treated With Placebo in 905-CL-076 | Adolescents Treated With Solifenacin in 905-CL-076
Started | 61 | 58 | 14 | 15
Safety Analysis Set (SAF) (SAF consisted of all participants with at least 1 dose of open-label solifenacin and safety data.) | 61 | 57 | 14 | 15
Full Analysis Set (FAS) (FAS consisted of all participants with at least 1 dose of open-label solifenacin and efficacy data.) | 60 | 57 | 14 | 15
Completed | 53 | 46 | 12 | 11
Not Completed | 8 | 12 | 2 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Adverse Event | 6 | 7 | 2 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — No Treatment Needed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is Safety Analysis Set (SAF), which consisted of all participants who received at least 1 dose of open-label solifenacin and had any safety data reported after the first dose of open-label solifenacin. The baseline values measured for study 905-CL-076 were used as the baseline values for the present study.
Groups:
- Adolescents Treated With Solifenacin in 905-CL-076: Male and female adolescents aged 12 to less than 18 years old who received solifenacin in Study 905-CL-076 and received open-label solifenacin once daily in this study. The mean time on study drug in this study was 240.1 days in adolescents.
- Total: Total of all reporting groups
Arm/Group | Children Treated With Placebo in 905-CL-076 | Children Treated With Solifenacin in 905-CL-076 | Adolescents Treated With Placebo in 905-CL-076 | Adolescents Treated With Solifenacin in 905-CL-076 | Total
Number analyzed (Participants) | 61 | 57 | 14 | 15 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The row for children only includes data for children. The row for adolescents only includes data for adolescents.
  Years
    Children: number analyzed (Participants) | 61 | 57 | 0 | 0 | 118
    Children | 7.2 (1.6) | 7.5 (1.5) |  |  | 7.3 (1.6)
    Adolescents: number analyzed (Participants) | 0 | 0 | 14 | 15 | 29
    Adolescents |  |  | 13.9 (1.6) | 14.5 (1.8) | 14.2 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 13 | 11 | 85
  Male | 34 | 23 | 1 | 4 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 2 | 1 | 17
  Not Hispanic or Latino | 54 | 50 | 12 | 14 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 1 | 0 | 7
  Asian | 4 | 5 | 1 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 2 | 7
  White | 49 | 47 | 11 | 12 | 119
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With and Severity of Treatment-Emergent Adverse Events (TEAEs)
Description: The investigator assessed the severity of AEs, including abnormal clinical laboratory values, electrocardiogram (ECG), vital signs, as follows:
  Mild: No disruption of normal daily activities; Moderate: Affect normal daily activities; Severe: Inability to perform daily activities. In participants treated with placebo in Study 905-CL-076, a TEAE was defined as an AE that started/worsened after the first dose of open-label solifenacin in Study 905-CL-077 up to 7 days after the last dose of solifenacin. In participants treated with solifenacin in Study 905-CL-076, a TEAE was defined as an AE that started/worsened after the first dose of double-blind solifenacin in Study 905-CL-076 up to 7 days after last dose of open-label solifenacin in Study 905-CL-077.
Time Frame: From first dose of solifenacin (in Study 905-CL-076 or in current study) up to 7 days after last dose of open-label solifenacin (41 weeks for participants who received placebo in 076 and 53 weeks for those who received solifenacin in 076).
Population: Safety Analysis Set (SAF). Participants who received placebo and participants who received solifenacin in Study 905-CL-076 are combined for analyses of efficacy and safety in this study.
Measure: Count of Participants; unit: Participants
Groups:
- Children (Aged 5 to Less Than 12 Years): Children aged 5 to less than 12 years old with OAB who received placebo or solifenacin in 905-CL-076, received a weight-based dose of open-label solifenacin oral suspension once daily for 40 weeks in this study. At the start of the 12-week titration period, the dose was adjusted according to the weight of the participant in order to deliver a plasma drug exposure equivalent to the 2.5 mg, 5 mg, 7.5 mg and 10 mg once daily oral tablet dose of solifenacin in adults.
- Adolescents (Aged 12 to Less Than 18 Years): Adolescents aged 12 to less than 18 years old with OAB who received placebo or solifenacin in 905-CL-076, received a weight-based dose of open-label solifenacin oral suspension once daily for 40 weeks in this study. At the start of the 12-week titration period, the dose was adjusted according to the weight of the participant in order to deliver a plasma drug exposure equivalent to the 2.5 mg, 5 mg, 7.5 mg and 10 mg once daily oral tablet dose of solifenacin in adults.
Arm/Group | Children (Aged 5 to Less Than 12 Years) | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 118 | 29
Participants
  TEAE - Mild | 72 | 10
  TEAE - Moderate | 20 | 8
  TEAE - Severe | 1 | 2
  Any TEAE | 93 | 20
  Drug-related TEAEs | 41 | 11
  Deaths | 0 | 0
  Serious TEAEs | 1 | 1
  Drug-related serious TEAEs | 0 | 0
  TEAEs leading to discontinuation | 12 | 5
  Drug related TEAEs leading to permanent discont. | 12 | 4

2. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours
Description: The mean number of incontinence episodes was based on 7-day diary data completed by participants prior to each visit from the start of 905-CL-076 to the end of 905-CL-077. An Incontinence episode is defined as an episode with any involuntary loss of urine. Data are reported by duration of solifenacin treatment based on the number of days from the date of first dose of solifenacin in either study 905-CL-076 or 905-CL-077 up to and including the study visit. Using equivalent treatment duration periods, data were combined for participants who received placebo and solifenacin in study 905-CL-076 within each age group.
Time Frame: Baseline (of 905-CL-076 study) and after 3, 6, 9, 12, 24, 40, and 52 weeks of solifenacin treatment
Population: Full Analysis Set (FAS) consisted of participants received at least one dose of open-label solifenacin and at least one of the efficacy variables with a valid baseline value and valid post-baseline data from diary completed after first dose of open-label solifencacin. Participants with available data at each time point are included in the analysis.
Measure: Mean (Standard Error); unit: incontinence episodes
Arm/Group | Children (Aged 5 to Less Than 12 Years) | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 117 | 29
incontinence episodes
  3 weeks solifenacin treatment: number analyzed (Participants) | 114 | 28
  3 weeks solifenacin treatment | -0.92 (0.18) | -1.05 (0.34)
  6 weeks solifenacin treatment: number analyzed (Participants) | 116 | 26
  6 weeks solifenacin treatment | -1.11 (0.17) | -1.40 (0.33)
  9 weeks solifenacin treatment: number analyzed (Participants) | 115 | 29
  9 weeks solifenacin treatment | -1.28 (0.19) | -1.48 (0.38)
  12 weeks solifenacin treatment: number analyzed (Participants) | 111 | 29
  12 weeks solifenacin treatment | -1.39 (0.20) | -1.66 (0.39)
  24 weeks solifenacin treatment: number analyzed (Participants) | 108 | 27
  24 weeks solifenacin treatment | -1.61 (0.19) | -1.73 (0.39)
  40 weeks solifenacin treatment: number analyzed (Participants) | 97 | 23
  40 weeks solifenacin treatment | -1.66 (0.23) | -1.49 (0.36)
  52 weeks solifenacin treatment: number analyzed (Participants) | 44 | 11
  52 weeks solifenacin treatment | -1.56 (0.22) | -1.34 (0.38)
Statistical Analysis 1: Comparison: Children (Aged 5 to Less Than 12 Years); Repeated measures ANCOVA (analysis of covariance) was used in this analysis, which included double-blind and/or open-label solifenacin treatment duration, gender, geographic region and randomized treatment group in Study 905-CL-076 as fixed effects, baseline as a covariate and "duration" repeated within participant; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = -0.95, 95% CI 2-sided [-1.19 to -0.71], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = -1.11, 95% CI 2-sided [-1.34 to -0.88], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = -1.26, 95% CI 2-sided [-1.53 to -1.00], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = -1.39, 95% CI 2-sided [-1.63 to -1.16], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = -1.54, 95% CI 2-sided [-1.76 to -1.32], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = -1.56, 95% CI 2-sided [-1.81 to -1.31], Standard Error of Mean 0.13
Statistical Analysis 7: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = -1.93, 95% CI 2-sided [-2.19 to -1.67], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = -0.93, 95% CI 2-sided [-1.62 to -0.23], Standard Error of Mean 0.35
Statistical Analysis 9: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = -1.38, 95% CI 2-sided [-2.09 to -0.68], Standard Error of Mean 0.36
Statistical Analysis 10: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = -1.40, 95% CI 2-sided [-2.09 to -0.70], Standard Error of Mean 0.35
Statistical Analysis 11: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = -1.58, 95% CI 2-sided [-2.27 to -0.88], Standard Error of Mean 0.35
Statistical Analysis 12: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = -1.80, 95% CI 2-sided [-2.50 to -1.10], Standard Error of Mean 0.35
Statistical Analysis 13: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = -1.57, 95% CI 2-sided [-2.29 to -0.85], Standard Error of Mean 0.36
Statistical Analysis 14: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = -2.00, 95% CI 2-sided [-2.83 to -1.17], Standard Error of Mean 0.42

3. Secondary Outcome: Change From Baseline in Number of Dry (Incontinence-Free) Days Per 7 Days
Description: The number of dry (incontinence-free) days was based on 7-day diary data completed by participants prior to each visit from start of 905-C L-076 to end of 905-C L-077. An incontinence-free day is a day without any incontinence episodes. Data are reported by duration of solifenacin treatment based on the number of days from the date of first dose of solifenacin in either study 905-CL-076 or 905-CL-077 up to and including the study visit. Using equivalent treatment duration periods, data were combined for participants who received placebo and solifenacin in study 905-CL-076 within each age group.
Time Frame: Baseline (of 905-CL-076 study) and after 3, 6, 9, 12, 24, 40, and 52 weeks of solifenacin treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: days
Arm/Group | Children (Aged 5 to Less Than 12 Years) | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 117 | 29
days
  3 weeks solifenacin treatment: number analyzed (Participants) | 114 | 28
  3 weeks solifenacin treatment | 1.17 (0.16) | 1.69 (0.53)
  6 weeks solifenacin treatment: number analyzed (Participants) | 116 | 26
  6 weeks solifenacin treatment | 1.28 (0.19) | 2.21 (0.56)
  9 weeks solifenacin treatment: number analyzed (Participants) | 115 | 29
  9 weeks solifenacin treatment | 1.59 (0.21) | 1.94 (0.50)
  12 weeks solifenacin treatment: number analyzed (Participants) | 111 | 29
  12 weeks solifenacin treatment | 1.60 (0.21) | 2.89 (0.51)
  24 weeks solifenacin treatment: number analyzed (Participants) | 108 | 27
  24 weeks solifenacin treatment | 2.09 (0.22) | 3.19 (0.51)
  40 weeks solifenacin treatment: number analyzed (Participants) | 97 | 23
  40 weeks solifenacin treatment | 2.15 (0.25) | 2.71 (0.59)
  52 weeks solifenacin treatment: number analyzed (Participants) | 44 | 11
  52 weeks solifenacin treatment | 2.57 (0.40) | 3.27 (0.73)
Statistical Analysis 1: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = 1.35, 95% CI 2-sided [0.97 to 1.73], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = 1.43, 95% CI 2-sided [1.02 to 1.83], Standard Error of Mean 0.20
Statistical Analysis 3: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = 1.72, 95% CI 2-sided [1.27 to 2.16], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = 1.80, 95% CI 2-sided [1.36 to 2.24], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = 2.21, 95% CI 2-sided [1.74 to 2.67], Standard Error of Mean 0.23
Statistical Analysis 6: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = 2.28, 95% CI 2-sided [1.79 to 2.77], Standard Error of Mean 0.25
Statistical Analysis 7: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = 2.84, 95% CI 2-sided [2.19 to 3.49], Standard Error of Mean 0.33
Statistical Analysis 8: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = 1.53, 95% CI 2-sided [0.17 to 2.89], Standard Error of Mean 0.69
Statistical Analysis 9: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = 1.90, 95% CI 2-sided [0.52 to 3.27], Standard Error of Mean 0.70
Statistical Analysis 10: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = 1.75, 95% CI 2-sided [0.39 to 3.10], Standard Error of Mean 0.69
Statistical Analysis 11: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = 2.69, 95% CI 2-sided [1.34 to 4.05], Standard Error of Mean 0.69
Statistical Analysis 12: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = 3.07, 95% CI 2-sided [1.70 to 4.43], Standard Error of Mean 0.69
Statistical Analysis 13: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = 2.45, 95% CI 2-sided [1.05 to 3.85], Standard Error of Mean 0.71
Statistical Analysis 14: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = 3.93, 95% CI 2-sided [2.34 to 5.53], Standard Error of Mean 0.81

4. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours
Description: The mean number of micturitions (urinations) was based on 7-day diary data completed by participants prior to each visit from start of 905-CL-076 to end of 905-CL-077. Data are reported by duration of solifenacin treatment based on the number of days from the date of first dose of solifenacin in either study 905-CL-076 or 905-CL-077 up to and including the study visit. Using equivalent treatment duration periods, data were combined for participants who received placebo and solifenacin in study 905-CL-076 within each age group.
Time Frame: Baseline (of 905-CL-076 study) and after 3, 6, 9, 12, 24, 40, and 52 weeks of solifenacin treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: micturitions
Arm/Group | Children (Aged 5 to Less Than 12 Years) | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 117 | 29
micturitions
  3 weeks solifenacin treatment: number analyzed (Participants) | 114 | 28
  3 weeks solifenacin treatment | -0.78 (0.18) | -1.29 (0.39)
  6 weeks solifenacin treatment: number analyzed (Participants) | 116 | 26
  6 weeks solifenacin treatment | -0.96 (0.20) | -1.38 (0.63)
  9 weeks solifenacin treatment: number analyzed (Participants) | 115 | 29
  9 weeks solifenacin treatment | -1.15 (0.20) | -1.15 (0.61)
  12 weeks solifenacin treatment: number analyzed (Participants) | 111 | 29
  12 weeks solifenacin treatment | -1.09 (0.21) | -1.24 (0.49)
  24 weeks solifenacin treatment: number analyzed (Participants) | 108 | 27
  24 weeks solifenacin treatment | -1.42 (0.21) | -1.01 (0.49)
  40 weeks solifenacin treatment: number analyzed (Participants) | 97 | 23
  40 weeks solifenacin treatment | -1.43 (0.24) | -1.39 (0.75)
  52 weeks solifenacin treatment: number analyzed (Participants) | 44 | 11
  52 weeks solifenacin treatment | -1.80 (0.43) | -0.81 (0.34)
Statistical Analysis 1: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = -0.98, 95% CI 2-sided [-1.27 to -0.69], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = -1.15, 95% CI 2-sided [-1.44 to -0.86], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = -1.31, 95% CI 2-sided [-1.60 to -1.02], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = -1.22, 95% CI 2-sided [-1.51 to -0.93], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = -1.50, 95% CI 2-sided [-1.80 to -1.21], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = -1.52, 95% CI 2-sided [-1.83 to -1.22], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Children (Aged 5 to Less Than 12 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = -1.83, 95% CI 2-sided [-2.22 to -1.43], Standard Error of Mean 0.20
Statistical Analysis 8: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = -0.93, 95% CI 2-sided [-1.73 to -0.13], Standard Error of Mean 0.39
Statistical Analysis 9: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = -0.94, 95% CI 2-sided [-1.48 to -0.40], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = -0.81, 95% CI 2-sided [-1.46 to -0.17], Standard Error of Mean 0.31
Statistical Analysis 11: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = -0.91, 95% CI 2-sided [-1.53 to -0.28], Standard Error of Mean 0.30
Statistical Analysis 12: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = -0.71, 95% CI 2-sided [-1.80 to -0.38], Standard Error of Mean 0.52
Statistical Analysis 13: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = -1.18, 95% CI 2-sided [-1.92 to -0.44], Standard Error of Mean 0.36
Statistical Analysis 14: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = -1.79, 95% CI 2-sided [-2.59 to -1.00], Standard Error of Mean 0.38

5. Secondary Outcome: Change From Baseline in Mean Number of Grade 3 or 4 Urgency Episodes Per 24 Hours in Adolescents
Description: Adolescent participants were also asked to record urgencies for at least 2 of the 7 diary days using the Perception of Intensity of Urgency Scale (PPIUS): (0 - no urgency, 1 - mild urgency, 2 - moderate urgency, 3 - severe urgency, 4 - urge incontinence). This data is based on 7-day diary data completed by participants prior to each visit from the start of 905-CL-076 to the end of 905-CL-077. Data are reported by duration of solifenacin treatment based on the number of days from the date of first dose of solifenacin in either study 905-CL-076 or 905-CL-077 up to and including the study visit. Using equivalent treatment duration periods, data were combined for participants who received placebo and solifenacin in study 905-CL-076 within each age group.
Time Frame: Baseline (of 905-CL-076 study) and after 3, 6, 9, 12, 24, 40, and 52 weeks of solifenacin treatment
Population: as for outcome 2
Measure: Mean (Standard Error); unit: urgency episodes
Arm/Group | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 29
urgency episodes
  3 weeks solifenacin treatment: number analyzed (Participants) | 27
  3 weeks solifenacin treatment | -0.79 (0.26)
  6 weeks solifenacin treatment: number analyzed (Participants) | 25
  6 weeks solifenacin treatment | -1.36 (0.53)
  9 weeks solifenacin treatment: number analyzed (Participants) | 27
  9 weeks solifenacin treatment | -1.15 (0.54)
  12 weeks solifenacin treatment: number analyzed (Participants) | 28
  12 weeks solifenacin treatment | -1.31 (0.38)
  24weeks solifenacin treatment: number analyzed (Participants) | 26
  24weeks solifenacin treatment | -1.11 (0.47)
  40 weeks solifenacin treatment: number analyzed (Participants) | 22
  40 weeks solifenacin treatment | -2.18 (0.81)
  52 weeks solifenacin treatment: number analyzed (Participants) | 10
  52 weeks solifenacin treatment | -1.87 (0.44)
Statistical Analysis 1: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 3 weeks; Adjusted change from baseline = -0.74, 95% CI 2-sided [-1.65 to 0.17], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 6 weeks; Adjusted change from baseline = -1.30, 95% CI 2-sided [-2.23 to -0.36], Standard Error of Mean 0.47
Statistical Analysis 3: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 9 weeks; Adjusted change from baseline = -1.14, 95% CI 2-sided [-2.06 to -0.22], Standard Error of Mean 0.47
Statistical Analysis 4: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 12 weeks; Adjusted change from baseline = -1.28, 95% CI 2-sided [-2.18 to -0.38], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 24 weeks; Adjusted change from baseline = -1.04, 95% CI 2-sided [-1.95 to -0.12], Standard Error of Mean 0.46
Statistical Analysis 6: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 40 weeks; Adjusted change from baseline = -1.96, 95% CI 2-sided [-2.93 to -1.00], Standard Error of Mean 0.49
Statistical Analysis 7: Comparison: Adolescents (Aged 12 to Less Than 18 Years); [analysis description as in outcome 2, analysis 1]; Test type: Other; Repeated Measures ANCOVA; Duration of solifenacin treatment: 52 weeks; Adjusted change from baseline = -2.20, 95% CI 2-sided [-3.48 to -0.93], Standard Error of Mean 0.65

6. Secondary Outcome: Change From Baseline to Final Visit in Postvoid Residual (PVR) Volume
Description: PVR volume was assessed by ultrasonography or bladder scan during 905-CL-076 and 905-CL-077. The value reported is the last PVR volume value after first dose of solifenacin up to 52 weeks.
Time Frame: Baseline (of 905-CL-076 study) to final Visit (the most recent value after first dose of solifenacin up to 40 weeks for participants who received placebo in 076 and 52 weeks for those who received solifenacin in 076.)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Children (Aged 5 to Less Than 12 Years) | Adolescents (Aged 12 to Less Than 18 Years)
Number analyzed (Participants) | 118 | 29
mL | 1.3 (11.9) | 0.7 (8.8)

ADVERSE EVENTS:
Time Frame: From first dose of solifenacin (in Study 905-CL-076 or in current study) up to 7 days after last dose of open-label solifenacin (41 weeks for participants who received placebo in 076 and 53 weeks for those who received solifenacin in 076).
Description: (1) For participants who received placebo in 905-CL-076, a TEAE was defined as any AE that started or worsened after the first dose of open-label solifenacin in 905-CL-077 and up to 7 days after the last dose of open-label solifenacin; (2) For subjects who received solifenacin in 905-CL-076, a TEAE is defined as any AE that started or worsened after the first dose of double-blind solifenacin in 905-CL-076 and up to 7 days after the last dose of open-label solifenacin.
Groups:
- Children (Aged 5 to Less Than 12 Years: Children aged 5 to less than 12 years old with OAB who received placebo or solifenacin in 905-CL-076, received a weight-based dose of open-label solifenacin oral suspension once daily for 40 weeks in this study. At the start of the 12-week titration period, the dose was adjusted according to the weight of the participant in order to deliver a plasma drug exposure equivalent to the 2.5 mg, 5 mg, 7.5 mg and 10 mg once daily oral tablet dose of solifenacin in adults.
Arm/Group | Children (Aged 5 to Less Than 12 Years | Adolescents (Aged 12 to Less Than 18 Years)
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/118 | 1/29
Other Adverse Events (participants affected / at risk) | 70/118 | 16/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children (Aged 5 to Less Than 12 Years (N=118) | Adolescents (Aged 12 to Less Than 18 Years) (N=29)
Gastroenteritis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Children (Aged 5 to Less Than 12 Years (N=118) | Adolescents (Aged 12 to Less Than 18 Years) (N=29)
Electrocardiogram QT prolonged (Investigations) | 10 | 4
Seasonal allergy (Immune system disorders) | 1 | 2
Headache (Nervous system disorders) | 16 | 1
Pyrexia (General disorders) | 9 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 16 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Escherichia urinary tract infection (Infections and infestations) | 7 | 2
Gastroenteritis (Infections and infestations) | 11 | 2
Nasopharyngitis (Infections and infestations) | 16 | 4
Urinary tract infection (Infections and infestations) | 6 | 2
Influenza (Infections and infestations) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 90 days prior to publication for review and comment. Sponsor may delay the publication temporarily to seek patent protection or permanently withhold the publication.